CLINICAL TRIAL: NCT06228768
Title: Acupressure for Aromatase Inhibitor-Associated Musculoskeletal Symptoms in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UMCC 2023.084; HUM00241228 (Other: University of Michigan); BCRF-23-206 (Other Grant/Funding Number: Breast Cancer Research Foundation)
Record Dates: First submitted 2024-01-16; First posted 2024-01-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Postmenopausal; Breast Cancer
Keywords: acupressure; arthralgia; aromatase inhibitor; joint pain; AIMSS
MeSH Terms: conditions — Breast Neoplasms; Arthralgia | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to two different sets of acupressure points
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both clinicians and participants will be blinded to study arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure Arm 1 (Other): There are 5 acupoints with 4 of the acupoints performed on both the left and right sides of the body. Each of the 9 acupoints will be stimulated for 3 minutes per point with the AcuWand giving a total treatment time of 27 minutes daily. The relaxation acupoints are unlisted in order to maintain blinding.
  Interventions: Other: Acupressure
- Acupressure Arm 2 (Other): There are 5 acupoints with 4 of the acupoints performed on both the left and right sides of the body. Each of the 9 acupoints will be stimulated for 3 minutes per point giving a total treatment time of 27 minutes daily. The acupoints are unlisted in order to maintain blinding.
  Interventions: Other: Acupressure

INTERVENTIONS:
Other: Acupressure — 9 acupoints will be stimulated for 3 minutes per point
  Arms: Acupressure Arm 1
Other: Acupressure — 9 areas will be stimulated for 3 minutes per point
  Arms: Acupressure Arm 2

SUMMARY:
This is a randomized, double-blinded trial of self-acupressure to examine the effect of treatment on aromatase inhibitor (AI)-associated musculoskeletal symptoms (AIMSS) in postmenopausal women with breast cancer. Acupressure is similar to acupuncture, but uses pressure rather than needles to stimulate specific points on the body. Acupressure involves applying mild to moderate physical pressure using your fingers, or an assistive device, to these points to try to bring about a physiological change in your body, in this case relief from joint pain and stiffness. The investigators will also examine effects of acupressure on other symptoms that commonly develop in AI-treated patients. In addition, changes in stool microbiome with acupressure treatment will be examined in an exploratory way to obtain preliminary information about the effect of acupressure on the gut microbiome in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subject aged ≥ 18 years
* Taking the currently prescribed aromatase inhibitor therapy (anastrozole, exemestane, or letrozole) for adjuvant or palliative treatment of breast cancer or for chemoprevention for at least 3 weeks and no more than 2 years at the time of enrollment.
* Planning to take the same AI therapy for at least 12 weeks.
* New or worsening joint pain and/or myalgias since starting the AI therapy, with worst pain score of at least 4 out of 10 on the BPI over the 7 days prior to enrollment.
* Completion of radiation therapy, if given, for treatment of breast cancer.
* Completion of chemotherapy, if given. Concurrent use of LHRHa therapy, anti-HER2 therapy, bisphosphonate therapy, PARP inhibitor therapy, and CDK4/6 inhibitor therapy is permitted.
* Patients receiving treatment with NSAIDs, acetaminophen, opioids, duloxetine, cannabinoids, gabapentin, and/or pregabalin must have been taking a stable dose for at least 30 days prior to enrollment if they plan to continue the drug during study participation. If they do not plan to take the medication during study participation, they should stop the medication at least 7 days before initiation of study treatment.
* Able to self-complete questionnaires in English.
* Able to access WiFi/internet and willing to use an email account or download and use the MyDataHelps app.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Use of acupuncture or acupressure in the past year, or planned use of acupuncture during study participation.
* Use of systemic or transdermal estrogen during study participation.
* Planned surgery during the 12-week study period.
* Concurrent medical or arthritis disease such as painful bone metastases or active rheumatoid arthritis or inflammatory arthritis that could confound or interfere with evaluation of pain or efficacy. Patients with osteoarthritis and asymptomatic bone metastases are eligible.
* Patients with a prior or concurrent malignancy whose natural history or treatment, in the opinion of the treating investigator, has the potential to interfere with the safety or efficacy assessment of the investigational regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2025-11-16 (Actual)

PRIMARY OUTCOMES:
Change in joint pain | baseline and 12 weeks after intervention is started
  Range 0-10 after 12 weeks of intervention. Brief Pain Inventory (BPI) questionnaire will be used for this assessment. Comparison of baseline and 12 week assessment.

SECONDARY OUTCOMES:
Proportion of patients with at least a 2 point reduction in pain (worst) | baseline and 12 weeks after intervention is started
  The proportion of patients who have at least a 2-point reduction in worst pain from baseline to 12 weeks will be reported with the corresponding exact binomial confidence intervals in each treatment group. The proportions will be compared using a chi-square test for each outcome. Differences from baseline at each time point for worst pain will be summarized via mean and standard deviation. Linear models using generalized estimating equations will assess the change in worst pain over time between groups similar to the primary endpoint. Brief Pain Inventory (BPI) questionnaire will be used for this assessment.
Proportion of patients with at least a 2 point reduction in pain (average) | baseline and 12 weeks after intervention is started
  The proportion of patients who have at least a 2-point reduction in average pain from baseline to 12 weeks will be reported with the corresponding exact binomial confidence intervals in each treatment group. The proportions will be compared using a chi-square test for each outcome. Differences from baseline at each time point for worst pain will be summarized via mean and standard deviation. Linear models using generalized estimating equations will assess the change in average pain over time between groups similar to the primary endpoint. Brief Pain Inventory (BPI) questionnaire will be used for this assessment.
Difference from baseline for pain interference | baseline, 6 weeks and 12 weeks after intervention is started
  Brief Pain Inventory (BPI) questionnaire will be used for this assessment. Differences from baseline at each time point for pain interference (range 0-10) will be summarized via mean and standard deviation. Linear models using generalized estimating equations will assess the change in pain interference over time between groups similar to the primary endpoint.
Change in reported sleep disturbance | baseline, 6 weeks and 12 weeks after intervention is started
  PROMIS Profile 29- sleep disturbance [range 32-73.3]. Patient reported outcomes will be analyzed using linear models and generalized estimating equations with robust variance similar to the primary outcome.
Change in reported fatigue | baseline, 6 weeks and 12 weeks after intervention is started
  PROMIS Profile 29-fatigue [range 33.7-75.8]. Patient reported outcomes will be analyzed using linear models and generalized estimating equations with robust variance similar to the primary outcome.
Change in reported physical function | baseline, 6 weeks and 12 weeks after intervention is started
  PROMIS Profile 29 -physical function [range 22.5-57]. Patient reported outcomes will be analyzed using linear models and generalized estimating equations with robust variance similar to the primary outcome.
Change in anxiety | baseline, 6 weeks and 12 weeks after intervention is started
  PROMIS Profile 29-anxiety [range 40.3-81.6].Patient reported outcomes will be analyzed using linear models and generalized estimating equations with robust variance similar to the primary outcome.
Change in depression | baseline, 6 weeks and 12 weeks after intervention is started
  PROMIS Profile 29-depression [range 41-79.4]. Patient reported outcomes will be analyzed using linear models and generalized estimating equations with robust variance similar to the primary outcome.
Change in cognitive function | baseline, 6 weeks and 12 weeks after intervention is started
  PROMIS Profile 29-cognitive function [range 29.4-61.2]. Patient reported outcomes will be analyzed using linear models and generalized estimating equations with robust variance similar to the primary outcome.
Adherence to trial intervention (number of days completed) | 12 weeks after intervention is started
  Adherence will be calculated based on number of days acupressure is performed The proportion of participants who are fully adherent will be compared between groups using a chi-square test.
Adherence to trial intervention (number of minutes completed) | 12 weeks after intervention is started
  Adherence will be calculated based on number of minutes of acupressure performed each day. The proportion of participants who are fully adherent will be compared between groups using a chi-square test.
safety of the intervention through reported adverse events | 12 weeks after intervention is started
  collected using CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Norah Henry, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
participant demographics and patient-reported outcomes data will be available to researchers upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: researchers can request data once the primary analysis has been published
Access Criteria: deidentified data will be available to researchers upon reasonable request

REFERENCES:
- [Derived] Henry NL, Kidwell KM, Kozar S, Snyder S, Zick SM. Self-acupressure for patients with breast cancer experiencing aromatase inhibitor-associated musculoskeletal symptoms: Protocol for the AcuAIM randomized pilot trial. PLoS One. 2025 Jan 22;20(1):e0311044. doi: 10.1371/journal.pone.0311044. eCollection 2025. PMID 39841658
- See also: Related Info — https://UMHealthResearch.org/studies/HUM00241228